CLINICAL TRIAL: NCT02020460
Title: A Clinical Evaluation of Direct Dorsal Column Stimulation for the Management of Chronic, Medically Refractory Neuropathic Pain
Brief Title: Clinical Evaluation of Direct Dorsal Column Stimulation
Acronym: DDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: Pro00036722
Record Dates: First submitted 2013-12-11; First posted 2013-12-25 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2015-08

CONDITIONS: Failed Back Surgery Syndrome
Keywords: post-laminectomy pain syndrome,; refractory,; refractory chronic neuropathic pain,; failed back surgery syndrome.
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subdural trial lead (Active Comparator): SCS trial lead in the subdural space.
  Interventions: Device: Subdural trial lead
- Epidural trial lead (Active Comparator): SCS trial lead in the epidural space.
  Interventions: Device: Epidural trial lead

INTERVENTIONS:
Device: Subdural trial lead
  Arms: Subdural trial lead
Device: Epidural trial lead
  Arms: Epidural trial lead

SUMMARY:
The study will examine the feasibility of Direct Dorsal Column Stimulation using existing Stimulation Leads (Ad-Tech). Secondary endpoints will include pain relief, somatosensory evoked potentials (SSEPs), stimulator settings required, improvement in quality of life and use of pain medications.

DETAILED DESCRIPTION:
Please note: This phase I feasibility study did not meet the expected enrollment goal of 75. The study only enrolled 6 subjects and therefore no participant completed phase II of the trial described below.

The primary objective of this study is to test the hypothesis that direct dorsal column stimulation is safe in the treatment of medically refractory, chronic neuropathic pain. The study will examine the feasibility of Direct Dorsal Column Stimulation using existing Stimulation Leads (Ad-Tech). Secondary endpoints will include pain relief, somatosensory evoked potentials (SSEPs), stimulator settings required, improvement in quality of life and use of pain medications.

Design & procedures This study is designed as a prospective, controlled exploratory study for an acute duration SCS trial system implantation. We will quantify perception of pain and stimulation-evoked paresthesias in response to both epidural and subdural direct dorsal column SCS. Additionally, we will measure the effects of both SCS modalities on somatosensory evoked potentials (SSEPs), patient quality of life, and satisfaction with treatment.

The normal clinical course of SCS for chronic pain includes a trial period of 3-30 days during which test stimulation is delivered via temporarily implanted epidural electrodes with an external percutaneous stimulation device. These electrodes are removed at the end of the trial period and, following a successful trial, a permanent set of electrodes and stimulation device are implanted at a later date. Subjects for this study will be recruited from patients planning to undergo percutaneous trial or paddle lead SCS implantation under the care of Dr. Nandan Lad at Duke University Medical Center.

Those subjects who a) have post-laminectomy pain syndrome and are considered good candidates for SCS trials, b) previously had successful SCS but have become refractory c) did not have adequate coverage during a prior SCS trial, or d) have been deemed refractory to all other treatments and would otherwise receive an intrathecal catheter/pump for chronic narcotics administration will be considered for participation.

Subjects recruited to this study will provide written informed consent prior to undergoing any research procedures (see "Selection of Subjects" below). Following consent and prior to surgery, we will record subject demographics and pain history, including age, sex, pain etiology, and history of prior pain-related surgeries. Subjects will then complete baseline assessments of pain using the revised short-form McGill Pain Questionnaire (SF-MPQ-2) and long form Brief Pain Inventory (BPI). Baseline measures for quality of life and global function will be measured with the EQ-5D-5L descriptive system and revised Self Assessment of Treatment (SAT) questionnaire, respectively.

After baseline measures have been recorded, the research study will be conducted in two phases. Study Phase I will occur during SCS implant surgery. First, an epidural trial SCS lead will be placed in accordance with the normal standard of care for this procedure. Next, a test stimulator (Cadwell ES-5) will be connected to the test lead and intraoperative test stimulation will be delivered for up to 30 minutes to determine the effect of spinal level, amplitude, frequency, pulse width on direct dorsal column stimulation. Sensation thresholds and paresthesia strength and coverage area will be recorded in response to these changes in stimulation parameters. SSEPs will be recorded throughout the procedure (Cadwell Cascade Elite IONM System). These will be recorded using needle electrodes placed on the tibial nerve and the scalp. Next, an Ad-tech subdural trial lead will be inserted in the standard fashion, similar to a standard lumbar drain catheter, and will be connected to the test stimulator. Test stimulation and quantification of responses will be repeated for up to an additional 30 minutes. The test stimulator will be disconnected once test stimulation is complete, and the surgery will continue per the normal standard of care to secure the two trial leads in place for post-operative percutaneous trial SCS.

Successful SCS trial lead placement is typically defined as at least 50% reduction in pain or adequate paresthesia coverage in the painful areas and the same threshold will be used for determining efficacy in both phases of the study. Subjects that do not meet either efficacy criterion will not be eligible to participate in the second phase of the study. The subdural trial electrode will be removed from these subjects, and they will continue with the normal clinical epidural SCS trial procedure.

Subjects entering Phase II of the study will be instructed to continue their usage of analgesic medications and other pain treatments as necessary, and will record any such use in the provided diary. This diary will also be used to query the subject for adverse events and side effects on a daily basis.

The second phase of the study will occur during the postoperative multi-day percutaneous SCS trial period. A hand-held trial stimulator typically used to deliver test stimulation during this trial period will be used to deliver stimulation for both standard care and the research study. A representative from St. Jude Medical (SJM) will work with each patient throughout the trial to program their system to its optimal setting, per the normal standard of care, but will not be involved in the collection of research data.

During the first half of study Phase II, trial SCS will be delivered to the subdural lead only (i.e. the epidural lead will be off). Methodological limitations prevent randomization of the order in which trial leads are activated in Phase II, so study staff will not be blinded to the location of the active SCS lead. However, subjects will not be told which trial lead is in use until the study is complete. The SJM representative will initially program the subdural trial lead on the day of surgery with standard stimulation settings. Subjects will assess their current pain intensity using a numeric rating scale (NRS) taken from the short-form BPI, item #6. Subjects will then be discharged from the hospital after receiving pain questionnaires and diaries to fill out over the next three days. On each of following two days, subjects will complete pain and quality of life ratings using the short from BPI, EQ-5D-5L descriptive system, and two NRS pain assessments; paresthesia coverage map and paresthesia quality ratings will also be completed to quantify sensory responses to SCS. On the third day following surgery, subjects will not complete NRS pain assessments, but will instead complete the SF-MPQ-2 and SAT in addition to the other ratings. This will conclude the first half of study Phase II.

The normal clinical course of trial stimulation will continue under the supervision of Dr. Lad and the SJM representative for up to 11 days to evaluate the efficacy of the trial SCS lead. Subjects will return to the Duke Spine Clinic (1B) at the end of this period for evaluation, x-ray imaging to confirm trial lead locations, and removal of the subdural trial lead. The epidural trial lead will then be activated, marking the beginning of the second half of study Phase II. All study procedures from the first half of Phase II will be repeated, this time using the epidural trial lead. Subjects will then continue normal clinical evaluation of the epidural trial lead with their care team, followed by removal of the epidural trial lead in the Duke Spine Clinic. The study team will review study participation with the subject and collect all remaining diaries at this time.

Description of Procedures performed:

The surgery is performed by the Principal Investigator, Dr. Nandan Lad MD, PhD.

Tuohy needle is percutaneously placed in the epidural space, using standard loss of resistance technique and a subdural stimulation lead is then passed and advanced under fluoroscopic guidance. The needle is then removed, and the lead is tested for stimulation and degree of pain relief. Figure of eight suture using 2.0 Silk is used to anchor to the skin.

Tuohy needle is then percutaneously placed in the lumbar subdural space, similar to a standard lumbar drain catheter insertion. An Ad-Tech lead is then passed and advanced under fluoroscopic guidance. The lead is tested for stimulation and degree of pain relief. The lead is anchored in place for post-operative percutaneous SCS trial (≤14 days). Figure of eight suture using 2.0 Silk is used to close the skin.

Trial leads will be removed by gently pulling and discarding the lead using the standard technique. All subjects will lay flat for 30 minutes to minimize the risk of low pressure headache following lead removal, consistent with standard practice for lumbar spinal catheters.

Selection of Subjects

It is anticipated that a total of 75 individuals will be studied. Subjects will be recruited from the Spine Clinic at Duke and overseen by Dr. Lad, respectively. Subjects will participate on a volunteer basis with informed consent approved by the Institutional Review Board of Duke University Medical Center. Apart from medically refractory chronic neuropathic pain, these individuals will be in good health. . The age range will be 18 years or older.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study must meet the following inclusion criteria:

1. Primary pain type-neuropathic with concordant neurologic findings
2. Subject age is 18 years or older;
3. Subjects who meet one of the following four criteria:

   1. diagnosed with medically refractory chronic neuropathic pain, post laminectomy pain syndrome or failed back surgery syndrome.
   2. previously had successful SCS, but gradually became refractory
   3. did not have adequate coverage during a prior SCS trial,
   4. been deemed refractory to all other treatments and would otherwise receive an intrathecal catheter/pump for chronic narcotics administration
4. Disease duration of at least 6 months with no lasting success with standard therapy and medications.
5. Mean pain intensity of at least 5 cm (or greater), measured on a visual analog scale from 0 (no pain) to 10 cm (severe pain) on a 10 cm line;
6. Psychological screening has been completed and the patient has been cleared by a psychologist or psychiatrist as a suitable SCS candidate;
7. Subject is willing to cooperate with the study requirements including compliance with the treatment regimen, the follow-up visit schedule and completion of the study diary;
8. Female candidates of childbearing potential must have a negative serum pregnancy test.
9. MRI or CT myelogram of the lumbar and thoracic spine (within 12 months prior to screening) rules out a pathology that might compromise SCS electrode placement or pathology, in addition to neural compression that might contribute to the subject's pain
10. Provide informed consent to participate in the study; -

Exclusion Criteria:

A subject will be excluded from participation in this study if they meet any one of the following criteria:

1. Pain attributed to: vascular disorder; musculoskeletal disorder; substance abuse or withdrawal; infection; disorder of homeostasis;
2. Subjects currently participating in another clinical trial;
3. Subject has an existing intrathecal drug pump
4. Active local or systemic infection
5. Unresolved issues of secondary gain (e.g., litigation)
6. Expected inability to adequately report treatment outcome
7. A concurrent clinically significant or disabling chronic pain problem or condition that is likely to confound evaluation of study endpoints (e.g., chronic migraine, significant arthritis of the hip associated with groin pain as primary complaint)
8. Radiographic evidence of frank instability (grossly mobile spondylolisthesis or abnormal subluxation) requiring fusion, calcific arachnoiditis, or severe thoracic or lumbar stenosis.
9. Subjects who have a condition that requires diathermy or repeat MRI's;
10. New medication for pain control has been initiated within 8 weeks prior to the initial baseline;
11. Female candidates of child bearing potential who are pregnant (confirmed by positive serum pregnancy test), not using adequate contraception as determined by the investigator, or nursing (lactating) a child;
12. Subject has a blood clotting disturbance or requires chronic anticoagulant drug therapy
13. The Investigator deems that the subject is not suitable for the study even if they meet all other inclusion/exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by interview and questionnaire | 3-5 days after Successful SCS trial lead placement defined as at least 50% reduction in pain or adequate paresthesia coverage in the painful areas.
  The subject will be asked to complete various questionnaires about their pain characteristics, consisting of pain rating scales and subjective recordings and ratings of stimulation intensity, duration, timing and location of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Nandan Lad, MD, PhD, Principal Investigator — DUMC
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States